CLINICAL TRIAL: NCT02558777
Title: Pilot Study of a Multicomponent Nurse Intervention to Reduce the Incidence and Severity of Delirium in Hospitalized Older Adults: MID-Nurse-P
Brief Title: Pilot Study of a Multicomponent Nurse Intervention to Reduce Delirium in Hospitalized Older Adults
Acronym: MID-Nurse-P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Complejo Hospitalario Universitario de Albacete (Other)
Responsible Party: Principal Investigator, Pedro Abizanda, MD,PhD, Complejo Hospitalario Universitario de Albacete
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MID-Nurse-P
Record Dates: First submitted 2015-07-28; First posted 2015-09-24 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Delirium
Keywords: Delirium; Pilot Study; Nurse intervention; Hospitalization
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): Multicomponent nurse-led intervention (orientation, sensorial deficit, sleep, mobilization, hydration, nutrition, drugs, elimination, oxygenation, pain)
  Interventions: Other: Multicomponent nurse-led intervention
- Control Group (No Intervention): Usual care

INTERVENTIONS:
Other: Multicomponent nurse-led intervention — Participants in the intervention group received the first intervention in the first 24 hours from admission, and thereafter daily until hospital discharge. The intervention was carried out exclusively by the "intervention nurses", and was composed of two main parts, being the first one a risk factor analysis, and the second one the intervention on the risk factors detected (orientation, sensorial deficit, sleep, mobilization, hydration, nutrition, drugs, elimination, oxygenation, pain). Furthermore, the intervention nurses identified the principal caregiver in the first 24 hours from admission, and provided an informative booklet about strategies and recommendations to prevent delirium incidence, including ambient strategies, orientation abilities, and identification of alert signs.
  Arms: Intervention Group

SUMMARY:
Objectives: To analyze if a multicomponent nurse-led intervention randomized clinical trial (MID-Nurse Study) is feasible (Pilot study), and can reduce the incidence, duration, and severity of delirium in hospitalized older adults in an AGU.

Design: Parallel-group Double-blind Randomized Clinical Trial (Pilot Study). Setting: AGU "Complejo Hospitalario Universitario from Albacete" (Albacete, Spain).

Participants: 50 patients ≥ 65 years hospitalized in the AGU (21 intervention group, 29 control group).

Interventions: After risk factor analysis, all participants in the intervention group (IG) received a daily multicomponent intervention (orientation, sensorial deficit, sleep, mobilization, hydration, nutrition, drugs, elimination, oxygenation, pain) by the intervention nurses. The control group (CG) received usual care.

Measurements: Delirium presence was determined daily with the Confusion Assessment Method (CAM), and delirium severity with the Delirium Rating Scale-Revised-98 (DRS). Mortality, days of hospitalization, use of physical restraint measures, and use of drugs for delirium control (neuroleptics and benzodiacepines) were also recorded.

DETAILED DESCRIPTION:
Parallel-group, double blind (evaluation and analysis), randomized clinical trial (pilot study). The design was based on recommendations for conducting pilot studies (Thabane 2010).

The main objective of the MID-Nurse (Randomized Clinical Trial) was to analyze if a multicomponent nurse-led intervention reduces the incidence, duration, and severity of delirium in hospitalized older adults in an Acute Geriatric Unit (AGU).

Specific objectives and evaluating criteria of the MID-Nurse-P (Pilot Study) were:

* Process: To determine the recruitment rate (criteria: at least 70% of the eligible patients can be recruited), the complete follow-up rate (criteria: at least 85% of the included participants complete the follow-up), and the adherence to intervention (criteria: at least 80% of the included participants receive every scheduled intervention).
* Resources: To assess capacity of the team and process time to conduct the trial. Criteria: Less than 10% of the participants can´t complete the intervention program due to study team problems, and daily time employed per participant is not longer than 30 minutes.
* Management: To analyze potential study personnel and data managing problems.
* Scientific: To estimate the intervention effect and the variance.

In the first 24 hours from admission, all the following data were collected by the evaluation nurses, once the informed consent was signed, and randomization performed by the principal investigator, who did not take part in the rest of the data collection and clinical intervention: Demographic data, Charlson comorbidity index, mean clinical diagnosis for admission, usually consumed drugs before admission, Barthel index, Holden´s FAC instrument, Pfeiffer´s Short Portable Mental Status Questionnaire, Reisberg´s Global Deterioration Scale, Dowton scale, pain with the visual analogical scale, and pressure ulcers risk with the Braden scale. Vital signs were determined on admission, including blood pressure, heart rate, temperature, hydration level, and oxygen saturation. Medical or nurse procedures were recorded, including bladder catheterization, nasogastric tube placement, venous or arterial access, blood sample acquisition, and other invasive procedures.

Blood sample was collected, and haemoglobin, leukocyte and neutrophil count, reactive C protein, sedimentation rate, glucose, urea, sodium, potassium, albumin, total proteins, cholesterol, thyroid stimulating hormone, transferrin, ferritin, total iron, folic acid, and B12 vitamin, were recorded.

After patient enrollment, all the patients received daily an evaluation of the Confusion Assessment Method scale (CAM) (Inouye 1990) by the evaluation nurses, in the afternoon. Prevalence of delirium throughout the follow-up was described, prevalence excluding the first day (to avoid bias of patients that were admitted with confusion), and incidence of delirium (new case across the follow-up, one patient could have more than 1 incident delirium). Number of days with delirium were also registered, and mean number of days with delirium was calculated for both groups.

In the case that the CAM was positive for delirium, patients also were evaluated with the Delirium Rating Scale-Revised-98 (DRS-R-98) (de Rooij 2006) to determine delirium severity. Total delirium severity was calculated by adding the severity of delirium during all days of hospitalization, and mean severity per day was calculated dividing the global severity per number of days with delirium.

Main outcome variables were the presence of delirium throughout the follow-up (dichotomic variable, yes/no), number of days with delirium during hospitalization (continuous variable), and total delirium severity (sum of DRS-R-98 during the complete follow-up).

Participants in the intervention group received the first intervention in the first 24 hours from admission, and thereafter daily until hospital discharge. Participants in the control group received usual medical and nurse care during all the hospitalization process. The intervention was carried out exclusively by the "intervention nurses", and was composed of two main parts, being the first one a risk factor analysis, and the second one the intervention on the risk factors detected (orientation, sensorial deficit, sleep, mobilization, hydration, nutrition, drugs, elimination, oxygenation, pain). Furthermore, the intervention nurses identified the principal caregiver in the first 24 hours from admission, and provided an informative booklet about strategies and recommendations to prevent delirium incidence, including ambient strategies, orientation abilities, and identification of alert signs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an age equal or older than 65 years
* Hospitalized at the Acute Geriatric Unit of the "Complejo Hospitalario Universitario of Albacete"
* Valid signed informed consent by the patient or legal representative.

Exclusion Criteria:

* Agonic situation
* Non-Spanish speaking
* Severe cognitive decline (Reisberg´s Global Deterioration Scale = 7)
* Patients sharing the same room with a previously included participant

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Delirium incidence (% participants) | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  Delirium incidence during hospitalization (% participants)

SECONDARY OUTCOMES:
Mean daily delirium severity (mean score Delirium Rating Scale-Revised-98) | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  Mean delirium severity per day with delirium (mean score Delirium Rating Scale-Revised-98)
Mortality (% of participants) | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  Mortality (% of participants)
Length of stay (days) | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  Length of hospitalization time (days)
Restraint measures (number of participants with these measures) | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  Use of restraint measures for delirium control (number of participants with these measures)
Drugs for delirium (% of participants using neuroleptics or benzodiazepines) | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  Use of drugs (neuroleptics or benzodiazepines) for delirium control (% of participants)
Delirium prevalence (% of participants) | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  Delirium prevalence during hospitalization (% of participants)
Delirium severity (sum of total Delirium Rating Scale-Revised-98 socres during hospitalization) | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  Delirium severity during hospitalization (sum of total Delirium Rating Scale-Revised-98 socres during hospitalization)
Recruitment rate (% of patients) | Up to five months
  % of the eligible patients recruited
Complete follow-up rate (% of participants) | Up to five months
  % of the included participants completing the follow-up
Adherence to intervention (% of participants) | Up to five months
  % of included participants receiving every scheduled intervention
Capacity of the team (% of participants) | Up to five months
  % of participants that can´t complete the intervention program due to study team problems
Process time (time in minutes) | Up to five months
  Daily time employed per participant for delivering the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Abizanda, MD,PhD, Principal Investigator — Complejo Hospitalario Universitario de Albacete (SESCAM)
Locations (1):
- Complejo Hospitalario Universitario de Albacete, Albacete, Albacete, Spain

REFERENCES:
- [Background] Inouye SK, Westendorp RG, Saczynski JS. Delirium in elderly people. Lancet. 2014 Mar 8;383(9920):911-22. doi: 10.1016/S0140-6736(13)60688-1. Epub 2013 Aug 28. PMID 23992774
- [Background] Hshieh TT, Yue J, Oh E, Puelle M, Dowal S, Travison T, Inouye SK. Effectiveness of multicomponent nonpharmacological delirium interventions: a meta-analysis. JAMA Intern Med. 2015 Apr;175(4):512-20. doi: 10.1001/jamainternmed.2014.7779. PMID 25643002
- [Background] Siddiqi N, Stockdale R, Britton AM, Holmes J. Interventions for preventing delirium in hospitalised patients. Cochrane Database Syst Rev. 2007 Apr 18;(2):CD005563. doi: 10.1002/14651858.CD005563.pub2. PMID 17443600
- [Background] Vidan MT, Sanchez E, Alonso M, Montero B, Ortiz J, Serra JA. An intervention integrated into daily clinical practice reduces the incidence of delirium during hospitalization in elderly patients. J Am Geriatr Soc. 2009 Nov;57(11):2029-36. doi: 10.1111/j.1532-5415.2009.02485.x. Epub 2009 Sep 15. PMID 19754498
- [Derived] Avendano-Cespedes A, Garcia-Cantos N, Gonzalez-Teruel Mdel M, Martinez-Garcia M, Villarreal-Bocanegra E, Oliver-Carbonell JL, Abizanda P. Pilot study of a preventive multicomponent nurse intervention to reduce the incidence and severity of delirium in hospitalized older adults: MID-Nurse-P. Maturitas. 2016 Apr;86:86-94. doi: 10.1016/j.maturitas.2016.02.002. Epub 2016 Feb 8. PMID 26921934